CLINICAL TRIAL: NCT02635581
Title: A DEXA Clinical Study to Evaluate the Osteointegrative Potential of Trabecular Titanium™
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Limacorporate S.p.a (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TT-01
Record Dates: First submitted 2015-12-15; First posted 2015-12-21 (Estimated); Last update posted 2016-03-02 (Estimated); Status verified 2016-03

CONDITIONS: Primary Total Hip Replacement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DELTA TT (Experimental)
  Interventions: Device: Delta TT acetabular cup

INTERVENTIONS:
Device: Delta TT acetabular cup

SUMMARY:
The purpose of this clinical trial is to evaluate the osteointegrative potential of the Trabecular TitaniumTM and to measure the pattern of changing in bone mineral density (BMD) around an uncemented acetabular cup, manufactured in Trabecular Titanium™ , during 60 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* BMI< 40 kg/m2
* Indication suitable to the implantation of Delta TT acetabular cup (First implant)
* Idiopathic osteoarthritis
* Avascular necrosis
* Post-traumatic arthritis
* Presence of sufficient periacetabular bone stock
* Ability to understand the investigation, cooperate with the investigational procedure and willing to return to the hospital for the required post-operative follow-ups
* Written informed consent

Exclusion Criteria:

* Patients found unsuitable for an implantation of Delta TT acetabular cup (Revision)
* Patients aged 76 or older
* Haemophilic disease
* Femur neck fracture
* Insulin Dependent Diabetes Mellitus (IDDM)
* Severe kidney failure (grade 4)
* Not responder Hypo- or Hyperthyroidism
* Paget's disease
* Tumours
* Active or suspicious infections
* Neurosensory deficits or neuromuscular diseases
* Severe and impairing vascular diseases
* Known incompatibility or allergy to products materials
* Woman with pregnancy or childbearing capacity or breast-feeding
* Subjects already enrolled in other clinical trials

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2008-12; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
The percentage change of the bone mineral density (BMD) around the acetabular cups with DEXA scan | From baseline to 5 year Follow-up

SECONDARY OUTCOMES:
Harris Hip Score (HHS) | From baseline to 5 year Follow-up
SF-36 score | From baseline to 5 year Follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Leo Massari, Principal Investigator — Azienda Ospedaliero-Universitaria di Ferrara, Arcispedale S. Anna
Locations (4):
- Italy (4):
  - Azienda Ospedaliero-Universitaria di Ferrara, Arcispedale S. Anna, Cona, Ferrara
  - Azienda Ospedaliero-Universitaria Città della Salute e della Scienza di Torino, Dipartimento di Ortopedia, Traumatologia e Riabilitazione, Ospedale CTO, Clinica II, Torino
  - Azienda Ospedaliero-Universitaria Città della Salute e della Scienza di Torino, Dipartimento di Ortopedia, Traumatologia e Riabilitazione, Ospedale CTO, Clinica I, Torino
  - Azienda Ospedaliero-Universitaria di Udine, Santa Maria della Misericordia, Udine